CLINICAL TRIAL: NCT00056550
Title: A Study to Assess the Incidence of Deep Vein Thrombosis (DVT) Following Prophylactic Intravenous Administration of Recombinant Human Antithrombin(rhAT) to Hereditary Antithrombin (AT) Deficient Patients in High Risk Situations.
Brief Title: Assess Incidence of Deep Vein Thrombosis(DVT)Following Administration of Recombinant Human Antithrombin (rhAT) to Hereditary Antithrombin(AT) Deficient Patients in High Risk Situations.
Acronym: rhAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: rEVO Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GTC AT III 01002
Record Dates: First submitted 2003-03-17; First posted 2003-03-18 (Estimated); Results first posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-08

CONDITIONS: Antithrombin Deficiency, Congenital
Keywords: Antithrombin Deficiency, Congenital; Antithrombin III Deficiency
MeSH Terms: conditions — Antithrombin III Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Recombinant Human Antithrombin (rhAT) infusion (Experimental): Loading and continuous infusion dose of rhAT to target and maintain an AT activity level > 80% and < 120% of normal.
  Interventions: Biological: Recombinant Human Antithrombin (rhAT)

INTERVENTIONS:
Biological: Recombinant Human Antithrombin (rhAT) — Biological/Vaccine: Recombinant human antithrombin(rhAT) Phase III clinical trial.
  Other Names: ATryn

SUMMARY:
Patients with hereditary antithrombin (AT) deficiency are at increased risk of venous thrombosis and pulmonary embolism, particularly during certain high risk procedures. The trial is focusing on patients with confirmed hereditary antithrombin deficiency who are undergoing a surgical procedure or induced/spontaneous labor and delivery. The study will test the safety and efficacy of recombinant human antithrombin (rhAT) by infusing rhAT prior to, during and following the period of risk or surgical procedure.

DETAILED DESCRIPTION:
Objectives :

1. Assess the safety of recombinant antithrombin (rhAT) in hereditary antithrombin (AT) deficient patients.
2. Assess the incidence of acute deep venous thrombosis(DVT) alone in patients with hereditary antithrombin (AT) deficiency in situations usually associated with a high risk for thromboembolic events after increasing and targeting functional AT activity at >80% and < 120% of normal by prophylactic IV administration of rhAT.
3. Clinically assess and determine the relevance of thromboembolic events other than acute DVT to rhAT administration.

ELIGIBILITY:
Inclusion Criteria:

* Have congenital AT deficiency with a personal or family history of venous thrombotic events.
* Have a history of congenital AT deficiency that includes 2 or more plasma AT activity levels of ≤ 60% normal.
* Are scheduled to have an elective procedure known to be associated with a high risk for occurrence of Deep Venous Thrombosis (DVT). This will include surgical patients or pregnant patients scheduled for cesarean section or delivery induction. In addition, hospitalized pregnant HD patients in active labor will be allowed into the study.
* Are at least 18 years of age, not exceeding 70 years of age.
* Have signed an informed consent form.
* Have a negative serum pregnancy test at screening and negative urine pregnancy test at baseline. This only applies to female surgical patients (not scheduled for cesarean section) of childbearing potential.
* Are able to comply with the requirements of the study protocol.

Exclusion Criteria:

* Patients who have a diagnosis of hereditary APC resistance, Factor V Leiden, Protein S or C deficiency, prothrombin gene mutation (G20210A), or acquired (lupus anticoagulant) thrombophilic disorder.
* Patients who are scheduled for a neurosurgical procedure or open-heart surgery.
* Patients who have an underlying medical condition, which in the opinion of the investigator, could complicate the assessment of the incidence of DVT.
* Patients who have a known allergy to goats or goat products.
* Patients who have participated in a study employing an investigational drug within 30 days of the start of their participation in the current trial.
* Patients using fondaparinux sodium, or are expected to be treated with fondaparinux sodium during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2002-12; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cambell Tait, MD, Principal Investigator — Royal Infirmary Glaskow
Locations (11):
- United States (2):
  - Marietta, Georgia
  - Charleston, South Carolina
- France (2):
  - Paris
  - Toulouse
- Germany (3):
  - Berlin
  - Hanover
  - Mannheim
- Milan, Italy
- Stockholm, Sweden
- United Kingdom (2):
  - Bristol
  - Manchester

REFERENCES:
- [Derived] DeJongh J, Frieling J, Lowry S, Drenth HJ. Pharmacokinetics of recombinant human antithrombin in delivery and surgery patients with hereditary antithrombin deficiency. Clin Appl Thromb Hemost. 2014 May;20(4):355-64. doi: 10.1177/1076029613516188. Epub 2013 Dec 11. PMID 24335249
- See also: Additional information on hereditary antithrombin disease — http://www.atiii.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GTC Biotherapeutics (GTC) established clinical trials sites in hospitals located in the United States and Europe. GTC provided an international clinical team to support site registration requirements once a patient was identified for treatment. The clinical trial started in December 2002 and completed in February 2004.
Pre-assignment Details: Fourteen hereditary antithrombin (AT) deficient patients were enrolled into the trial. The patients included surgical (N = 5) and delivery patients (N = 9) who were treated with recombinant human antithrombin (rhAT) replacement therapy.
Groups:
- Recombinant Human Antithrombin (rhAT) Infusion: Following a baseline evaluation phase hereditary antithrombin(AT)deficient patients scheduled for surgery, cesarean section or vaginal delivery were planned to be treated prophylactically with recombinant human antithrombin (rhAT). Dosing with recombinant human antithrombin (rhAT) was individualized with an initial intravenous loading dose, followed by a continuous intravenous infusion dose, intended to target and maintain antithrombin (AT) activity levels > 80% and < 120% of normal. The dosing objective for all study patients is maintenance of the AT activity at >80% and <120% of normal during the high risk period for thromboembolic events. Dosing and dose adjustments were based on the results of AT activity level determinations performed prior to and during the treatment.
Period: Overall Study
Arm/Group | Recombinant Human Antithrombin (rhAT) Infusion
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Recombinant Human Antithrombin (rhAT) Infusion: Following a baseline evaluation phase hereditary AT deficient patients(previously documented AT activity < or equal to 60% of normal)scheduled for surgery ,cesarean section or vaginal delivery were planned to be treated prophylactically with rhAT. Dosing with rhAT was to be individualized with an initial loading dose, followed by a continuous maintenance infusion dose, intended to increase and target antithrombin (AT) activity levels > 80% and < 120% of normal.
Arm/Group | Recombinant Human Antithrombin (rhAT) Infusion
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 36.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Europe | 12
  United States | 2
Prior history of venous thrombotic events [Number; unit: Participants] — Inclusion criteria states that patients had to have congenital antithrombin (AT) deficiency with a personal or family history of venous thrombotic events.
  Participants | 14
Antithrombin (AT) activity level < or equal to 60% [Number; unit: Participants] — Inclusion criteria states that the patients must have a history of congenital antithrombin (AT) deficiency that includes two or more plasma AT activity levels < or equal to 60% of normal
  Participants | 14

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Thromboembolic Events Acute Deep Venous Thrombosis (DVT) and/or Thromboembolic Events Other Than Acute Deep Vein Thrombosis (DVT).
Description: Observation for clinical signs and symptoms of thromboembolic events are evaluated for acute deep vein thrombosis (DVT) using duplex ultrasonography and/or other imaging tests to confirm clinical signs/symptoms. Duplex ultrasonography was performed at baseline, last day of dosing and day 7 (+ or -1 day).
Time Frame: Baseline, last day of dosing and day 7 (+ or - 1 day)
Population: 14 patients who received at least 1 dose of rhAT were included in the Safety population. During the central review of the duplex ultrasound, 1 delivery patient was diagnosed with a DVT at baseline, and was not evaluable for efficacy, the patient was excluded from the PP population.
Measure: Number; unit: participants
Groups:
- Recombinant Human Antithombin (rhAT) Infusion: Following a baseline evaluation phase hereditary antithrombin (AT) deficient patients scheduled for surgery, cesarean section or vaginal delivery were planned to be treated prophylactically with recombinant human antithrombin (rhAT). Dosing with rhAT was to be individualized with an initial loading dose, followed by a continuous maintenance infusion dose, intended to target and maintain antithrombin (AT) activity levels > 80% and < 120% of normal. The dosing objective for all study patients is maintenance of the AT activity at >80 and < 120% of normal during the high risk period for thromboembolic events. Dosing and dose adjustments will be based on the results of AT activity determinations performed prior to and during treatment.
Arm/Group | Recombinant Human Antithombin (rhAT) Infusion
Number analyzed (Participants) | 14
participants | 1

2. Secondary Outcome: Local Assessment of Thromboembolism by Physical Examination.
Description: The investigators evaluated patients for any clinical signs of thromboembolism by physical examination.
Time Frame: 30 days after last dose
Population: 14 patients were included in the trial and treated with rhAT.
Measure: Number; unit: Participants in study
Groups:
- Recombinant Human Antithrombin (rhAT) Infusion: Following a baseline evaluation phase hereditary AT deficient patients scheduled for surgery ,cesarean section or vaginal delivery were planned to be treated prophylactically with rhAT. Dosing with rhAT was to be individualized with an initial loading dose, followed by a continuous maintenance infusion dose, intended to target and maintain antithrombin (AT) activity levels > 80% and < 120% of normal.
Arm/Group | Recombinant Human Antithrombin (rhAT) Infusion
Number analyzed (Participants) | 14
Participants in study | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for duration of study up to 90 days post study drug administration.
Description: All 14 patients who received rhAT were evaluated for the occurrence of treatment-emergent AEs from the time of their initial bolus dose up to and including 30 days after administration of their last dose of rhAT and for the development of antibodies to rhAT out to 90 days following treatment.
Arm/Group | Recombinant Human Antithrombin (rhAT) Infusion
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human Antithrombin (rhAT) Infusion (N=14)
Fever (General disorders) | 1 (1)
Thrombophlebitis Deep (Vascular disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Hemorrhage NOS (Blood and lymphatic system disorders) | 1 (1)
Convulsions Grand Mal (Nervous system disorders) | 1 (1)
Fracture Trauma (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human Antithrombin (rhAT) Infusion (N=14)
Hypotension (Cardiac disorders) | 1 (5)
Post-operative pain (General disorders) | 1 (4)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Nausea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Infection (General disorders) | 1 (2)
Hematoma (Blood and lymphatic system disorders) | 1 (3)
Fever (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No